CLINICAL TRIAL: NCT06987370
Title: A Phase II Randomized Controlled Clinical Study on the Efficacy and Safety Evaluation of Radiotherapy Mode Based on SFRT and SCART Technologies for Bone Metastatic Malignant Tumors With Soft Tissue Formation
Brief Title: SFRT and SCART in Radiotherapy for Bone Metastases With Soft Tissue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Directorof Radiation Oncology Department, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2025-076-03
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-05

CONDITIONS: Bone Metastases in Subjects With Advanced Cancer
Keywords: bone metastases; bone metastases with soft tissue; SFRT; SCART

STUDY DESIGN:
Intervention Model Description: This study intends to recruit 90 patients with bone metastases with soft tissue formation and randomly assign them to the experimental group and the group in a ratio of 2:1. The experimental group will be treated with either Spatially Fractionated Radiotherapy (SFRT) or Stereotactic Central Adaptive Radiotherapy (SCART) for the bone metastatic lesions (8-12 Gy in 1 fraction for vertices/SCART- treatment volume in the soft tissue lesions followed by 25-40 Gy in 5 fractions for the whole bone metastatic lesions). The control group will receive conventional external radiotherapy with a dose of 30 Gy in 10 fractions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SFRT/SCART GROUP (Experimental): Stereotactic Central Ablative Radiotherapy (SCART):
  When using SCART to treat bone metastases with associated soft tissue components, the gross tumor volume (GTV) of the bone metastases must be accurately delineated according to the guidelines. The GTV are contracted to derive the SCART-Treatment Volume (STV). An initial dose of 8-12 Gy in a single fraction is delivered to the STV, followed by a dose of 25-40 Gy in 5 fractions to the clinical target volume (CTV).
  Spatially Fractionated Radiotherapy (SFRT):
  The GTV are reduced to form a "LATTICE" target area. Several vertices are uniformly contoured along the edges of the "LATTICE." A dose of 8-12 Gy in a single fraction is delivered to the vertices, followed by a dose of 25-40 Gy in 5 fractions to the CTV.
  Interventions: Radiation: SCART (Stereotactic Central Ablative Radiation Therapy ) /SFRT（Spatially Fractionated Radiation Therapy ）
- Conventional Radiotherapy (CRT) Group (Active Comparator): The conventional radiotherapy group, that is, the control group, delineated the target areas in accordance with the consensus guidelines on the definition of target volumes in spinal stereotactic radiosurgery by the International Spine Radiosurgery Consortium and other relevant guidelines according to the location of bone metastases, and administered conventional external beam radiotherapy with a dose of 30 Gy in 10 fractions to the bone metastasis lesions.
  Interventions: Radiation: Conventional Radiotherapy (CRT)

INTERVENTIONS:
Radiation: Conventional Radiotherapy (CRT) — The conventional radiotherapy group, that is, the control group, administering conventional external beam radiotherapy with a dose of 30 Gy in 10 fractions to the bone metastasis lesions.
  Other Names: CRT group
  Arms: Conventional Radiotherapy (CRT) Group
Radiation: SCART (Stereotactic Central Ablative Radiation Therapy ) /SFRT（Spatially Fractionated Radiation Therapy ） — Stereotactic Central Ablative Radiotherapy (SCART): When using SCART to treat bone metastases with associated soft tissue components, the gross tumor volume (GTV) of the bone metastases must be accurately delineated according to the guidelines. The GTV are contracted to derive the SCART-Treatment Volume (STV). An initial dose of 8-12 Gy in a single fraction is delivered to the STV, followed by a dose of 25-40 Gy in 5 fractions to the clinical target volume (CTV). Spatially Fractionated Radiation Therapy (SFRT): The GTV are reduced to form a "LATTICE" target area. Several vertices are uniformly contoured along the edges of the "LATTICE." A dose of 8-12 Gy in a single fraction is delivered to the vertices, followed by a dose of 25-40 Gy in 5 fractions to the CTV.
  Other Names: SCART (Stereotactic Core Ablative Radiation Therapy ) /SFRT（Spatially Fractionated Radiation Therapy ）; SCART/SFRT group
  Arms: SFRT/SCART GROUP

SUMMARY:
This is a randomized, controlled, prospective phase II, two-arm clinical study designed to evaluate the efficacy and safety of using either Spatially Fractionated Radiotherapy (SFRT) or Stereotactic Central Ablative Radiotherapy (SCART) for treating the soft tissue components of malignant bone metastases. The study plans to enroll 90 patients with bone metastases accompanied by soft tissue formation, who will be randomized in a 2:1 ratio to the SFRT/SCART group or the conventional radiotherapy (CRT) group.The primary endpoint is the objective response rate (ORR). Tumor response to treatment will be assessed every 12 weeks (±7 days) according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Secondary endpoints include pain relief rate, progression-free survival (PFS), and safety. In addition, adverse events (AEs) will be monitored throughout the study.

DETAILED DESCRIPTION:
Bone is a common site for tumor metastasis, with approximately 18.8 out of every 100,000 cancer patients diagnosed with bone metastases each year. Lung cancer, prostate cancer, and breast cancer are the most common primary tumor types leading to bone metastases. Currently, there is limited research on bone metastases accompanied by soft tissue formation. However, such formations have been observed in the majority of bone metastasis cases originating from solid tumors. Conventional radiotherapy regimens for bone metastases often show poor local control over the soft tissue component. Based on above undergrounds, this study is designed to be a random, controlled, prospective phase II, two-arm clinical study. Totally 90 patients with bone metastasis accompanied by soft issue formation will be enrolled and randomized in a 2:1 ratio to the Spatially Fractionated Radiotherapy (SFRT)/ Stereotactic Central Ablative Radiotherapy (SCART) group or the conventional radiotherapy (CRT) group with the primary endpoint being the objective response rate (ORR) of the target lesion at 3, 6, 9, and 12 months post-radiotherapy, assessed using RECIST 1.1. Secondary endpoints include pain relief rate, PFS and safety (per CTCAE v5.0). Eligibility criteria include patients aged 18-75 years, ECOG performance status ≤2, and an expected survival of ≥3 months. Those with secondary primary tumors, pathological fracture confirmed by CT or MRI, patients who received radiotherapy to the target lesion prior to enrollment or women who are pregnant or breastfeeding will be excluded. Comprehensive baseline assessments (imaging, pathology, laboratory tests) are conducted pretreatment, with weekly toxicity monitoring during treatment. Efficacy assessments consist of ORR of 3,6,9,12 months and tumor-related pain evaluation. During the course of radiotherapy, patient-reported pain is measured using the Numeric Rating Scale (NRS) every week. After the completion of radiotherapy, pain assessments are conducted every 6 weeks. Imaging evaluations are performed every 12 weeks after completion of radiotherapy and include high-resolution MRI, CT of bone metastatic sites. Statistical analysis assumes a one-sided α=0.05, β=0.8, anticipating an ORR of 90% for SFRT/SCART versus 66% for CRT. This study aims to evaluate the efficacy and safety of using either Spatially Fractionated Radiotherapy (SFRT) or Stereotactic Central Ablative Radiotherapy (SCART) for treating the bone metastases with soft tissue formation.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent form before implementing any trial-related procedures; 2. Male or female, aged 18 years or above and 75 years or below; 3. Have a histopathologically confirmed single primary tumor (patients with a pathological diagnosis of small cell carcinoma or undifferentiated carcinoma are excluded); 4. ECOG PS 0-2; 5. Have at least one target lesion: bone metastasis with a soft tissue mass confirmed by CT or MRI. The shortest diameter of the soft tissue is greater than 30mm; 6. The number of metastatic lesions is ≤ 5 and the number of metastatic organs is ≤ 3; 7. The expected survival time is ≥ 3 months; 8. The main organ functions are normal (within 14 days before enrollment), that is, the following criteria are met:

1. The blood routine examination criteria should meet:

   1. Hemoglobin (HB) ≥ 90g/L;
   2. Absolute neutrophil count (ANC) ≥ 1.5×10⁹/L;
   3. Platelet count (PLT) ≥ 75×10⁹/L;
2. There is no functional organic disease, and the following criteria should be met:

   1. When there is no liver metastasis, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5× ULN, serum total bilirubin ≤ 1.5× ULN, alkaline phosphatase (ALP) ≤ 3× ULN; when there is liver metastasis, ALT and AST ≤ 5× ULN, serum total bilirubin ≤ 3× ULN, and alkaline phosphatase (ALP) ≤ 5× ULN;
   2. Serum creatinine level Cr ≤ 1.5×ULN (if the serum creatinine is elevated, a 24-hour urine collection is required, except for those with a 24-hour creatinine clearance rate > 50ml/min);
   3. Urine protein < 2+. If the test strip result is ≥ 2+, the 24-hour urine protein must be < 2g, or the urine protein-to-creatinine ratio (UPC) must be < 2;
   4. International normalized ratio (INR) and activated partial thromboplastin time (APTT): ≤ 1.5×ULN;

Exclusion Criteria:

1. Pathological fracture confirmed by CT or MR.
2. Prior radiotherapy to the target lesion.
3. Pregnant or lactating women.
4. Acute infection or other serious underlying diseases.
5. Obvious history of neurological and mental diseases, including dementia that may affect the ability to understand and give informed consent.
6. History or evidence of diseases, treatments or abnormal laboratory test values that may interfere with the test results and prevent the subject from participating in the study throughout the whole process, or other situations that the researcher deems inappropriate for enrollment. The researcher believes that there are other potential risks that make the subject unsuitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 year
  Defined as the proportion of patients whose tumor size decreases (partial response) or disappears (complete response) after radiation based on RECIST 1.1. (CR, complete disappearance of the lesion) or partial response (PR, ≥30% reduction in lesion diameter sum) at 3, 6, 9, and 12 months post-radiotherapy, evaluated according to RECIST 1.1.

SECONDARY OUTCOMES:
The pain relief rate | 1 year
  The NRS score is used as an indicator of the treatment response. Complete remission is defined as the absence of pain three months after radiotherapy. Partial remission is defined as the pain score being at least 2 points lower than the initial score (or the daily dosage of narcotic drugs decreasing by more than 20%). The stable state is defined as the change in the pain score not exceeding 1 point (or the change in the daily dosage of narcotic drugs not exceeding 10%). A progressive response is defined as the pain score being at least 2 points higher than the initial score (or the daily dosage of narcotic drugs increasing by more than 20%).
Local control rate | 1 year
  Local control rate is defined as the time from the start of radiotherapy to either progression of the target lesion (assessed per RECIST 1.1 criteria) or patient death from any cause, whichever occurs first.
Adverse event incidence (Safety) | 1 year
  Treatment-related adverse events are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, Doctor, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunne EM, Sahgal A, Lo SS, Bergman A, Kosztyla R, Dea N, Chang EL, Chang UK, Chao ST, Faruqi S, Ghia AJ, Redmond KJ, Soltys SG, Liu MC. International consensus recommendations for target volume delineation specific to sacral metastases and spinal stereotactic body radiation therapy (SBRT). Radiother Oncol. 2020 Apr;145:21-29. doi: 10.1016/j.radonc.2019.11.026. Epub 2019 Dec 23. PMID 31874346
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Nguyen TK, Chin L, Sahgal A, Dagan R, Eppinga W, Guckenberger M, Kim JH, Lo SS, Redmond KJ, Siva S, Stish BJ, Chan R, Lawrence L, Lau A, Tseng CL. International Multi-institutional Patterns of Contouring Practice and Clinical Target Volume Recommendations for Stereotactic Body Radiation Therapy for Non-Spine Bone Metastases. Int J Radiat Oncol Biol Phys. 2022 Feb 1;112(2):351-360. doi: 10.1016/j.ijrobp.2021.09.004. Epub 2021 Sep 9. PMID 34509549
- [Background] Cox BW, Spratt DE, Lovelock M, Bilsky MH, Lis E, Ryu S, Sheehan J, Gerszten PC, Chang E, Gibbs I, Soltys S, Sahgal A, Deasy J, Flickinger J, Quader M, Mindea S, Yamada Y. International Spine Radiosurgery Consortium consensus guidelines for target volume definition in spinal stereotactic radiosurgery. Int J Radiat Oncol Biol Phys. 2012 Aug 1;83(5):e597-605. doi: 10.1016/j.ijrobp.2012.03.009. Epub 2012 May 19. PMID 22608954
- [Background] Wu X, Perez NC, Zheng Y, Li X, Jiang L, Amendola BE, Xu B, Mayr NA, Lu JJ, Hatoum GF, Zhang H, Chang SX, Griffin RJ, Guha C. The Technical and Clinical Implementation of LATTICE Radiation Therapy (LRT). Radiat Res. 2020 Dec 1;194(6):737-746. doi: 10.1667/RADE-20-00066.1. PMID 33064814
- [Background] Yang J, Lu Q, Qi W, Kolb RD, Wang L, Li Y, Li S, Lin Y, Liu J, Mourad W, MirkhaghaniHaghighi F, Slavisa T, Wu X, You WC, Yang E, Hanlon A, Zhu A, Yan W. Stereotactic central/core ablative radiation therapy: results of a phase I study of a novel strategy to treat bulky tumor. Front Oncol. 2024 May 24;14:1364627. doi: 10.3389/fonc.2024.1364627. eCollection 2024. PMID 38854732
- [Background] Jung IH, Yoon SM, Kwak J, Park JH, Song SY, Lee SW, Ahn SD, Choi EK, Kim JH. High-dose radiotherapy is associated with better local control of bone metastasis from hepatocellular carcinoma. Oncotarget. 2017 Feb 28;8(9):15182-15192. doi: 10.18632/oncotarget.14858. PMID 28146433
- [Derived] Kou Y, Xu K, Zhu K, Jiang S, Feng R, Dou X, Xu L, Zhang X, Shi F, Liu X, Gong Z, Yue J. Efficacy and safety evaluation of radiotherapy approach based on spatially fractionated radiotherapy and stereotactic core ablative radiation therapy technologies for bone metastatic malignant tumors with soft tissue formation: A randomized controlled phase II trial. Precis Radiat Oncol. 2025 Dec 19;9(4):260-265. doi: 10.1002/pro6.70036. eCollection 2025 Dec. PMID 41477287